CLINICAL TRIAL: NCT03263351
Title: Depression and Insulin Sensitivity in Adolescents
Brief Title: Depression & Insulin Sensitivity in Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Colorado State University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Center for Advancing Translational Sciences (NCATS) (NIH); Children's Hospital Colorado (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 4185; R01DK111604 (NIH)
Record Dates: First submitted 2017-08-24; First posted 2017-08-28 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Type2 Diabetes; Type 2 Diabetes Mellitus; Insulin Sensitivity; Insulin Resistance; Depression; Adolescent Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance; Depression; Pediatric Obesity

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled behavioral trial with two conditions - cognitive-behavioral therapy group or health education group - run in parallel.
Who Masked: Outcomes Assessor
Masking Description: Research staff who assess outcomes will be blinded to condition assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cognitive-behavioral therapy group (Experimental): Six-session cognitive-behavioral therapy group program designed as a prevention of depression intervention for adolescents at-risk for depression. The program is facilitated by a psychologist. Sessions are weekly for 1-hour.
  Interventions: Behavioral: Cognitive-behavioral therapy group
- Health education group (Active Comparator): Six-session health education group program designed as a health education curriculum for teenagers. The program is facilitated by a psychologist. Sessions are weekly for 1-hour.
  Interventions: Behavioral: Health education group

INTERVENTIONS:
Behavioral: Cognitive-behavioral therapy group — Psychoeducation on depression; cognitive restructuring of negative thoughts; engagement in pleasant activities; healthy rewards; stress and coping.
  Other Names: Blues Program
  Arms: Cognitive-behavioral therapy group
Behavioral: Health education group — Didactic health knowledge about interpersonal violence; basic nutrition guidance; sun safety; depression and signs of suicide; gang violence; substance use.
  Other Names: Hey-Durham
  Arms: Health education group

SUMMARY:
There has been a rise in type 2 diabetes (T2D) rates in adolescents, disproportionately in girls from disadvantaged racial/ethnic groups. This group of girls also is at heightened risk for depression, and depression and T2D are linked. Depressive symptoms are a risk factor for worsening of insulin sensitivity, one if the major precursors to T2D. In preliminary studies, the investigators found that a brief cognitive-behavioral therapy group decreased depressive symptoms and prevented worsening of insulin sensitivity in adolescent girls at-risk for T2D with moderate depressive symptoms. The aims of this study are: 1) to assess the efficacy of a cognitive-behavioral therapy depression group vs. a health education control group for improving insulin sensitivity and preserving insulin secretion in racially/ethnically diverse adolescent girls at-risk for T2D with moderate depressive symptoms over a 1-year follow-up; 2) to evaluate changes in eating, physical activity, and sleep as explanatory and 3) to test changes in cortisol factors as explanatory.

DETAILED DESCRIPTION:
There has been rapid escalation of type 2 diabetes (T2D) rates in adolescents. Early-onset T2D (<20y) typically shows a more aggressive course than adult-onset T2D and disproportionately affects girls from disadvantaged, racial/ethnic groups. This group of girls also is at heightened risk for depression, and depression and T2D are linked. Depressive symptoms often manifest in adolescence and are a prospective risk factor for worsening of insulin sensitivity, the major physiological precursor-in combination with deterioration of pancreatic β-cell capacity to secrete insulin-in the path to T2D. The effects of depression on poor insulin sensitivity remain even after accounting for adiposity. In theory, depressive symptoms may worsen insulin sensitivity through stress-induced behaviors (e.g., disinhibited eating, physical inactivity, sleep disturbance) and stress-induced physiological causal mechanisms (e.g., hypercortisolism). The central theme of this study is that intervening to reduce depressive symptoms in adolescents at-risk for T2D may offer an innovative, targeted approach to ameliorate insulin resistance and to, consequently, preserve β-cell function and lessen T2D risk. In preliminary data, the investigators found initial evidence that a 6-week cognitive-behavioral group decreased depressive symptoms and prevented worsening of insulin sensitivity 1 year later in overweight and obese girls with moderate depressive symptoms and a family history of T2D, in comparison to a 6-week health education control group. Directly extending these findings, the primary aims of this study are: 1) to assess the efficacy of a 6-week cognitive-behavioral depression group vs. a 6-week health education control group for improving insulin sensitivity and preserving β-cell function in racially/ethnically diverse adolescent girls at-risk for T2D with moderate depressive symptoms over a 1-year follow-up; 2) to evaluate changes in eating, physical activity, and sleep as behavioral explanatory mediators underlying the relationship between decreases in depressive symptoms and improvements in insulin sensitivity and β-cell function over 1 year and 3) to test changes in cortisol awakening response, diurnal cortisol rhythm, and total daily cortisol output as physiological mechanisms explaining the relationship between decreases in depressive symptoms and improvements in insulin sensitivity and β-cell function over 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age 12-17 years
* Body mass index (BMI) ≥85th percentile for age & sex
* Center for Epidemiologic Studies-Depression Scale (CES-D) >20
* English speaking
* ≥1 first- or second-degree family member with type 2 diabetes (T2D), prediabetes, or gestational diabetes
* Good general health

Exclusion Criteria:

* Pregnancy or breastfeeding
* Type 2 diabetes as indicated by fasting glucose≥126 mg/dL or 2-hour glucose>200 mg/dL or Hba1c>=6.5
* Medication affecting mood, weight, cortisol, or insulin sensitivity, including insulin sensitizers (e.g., metformin), anti-depressants, and stimulants
* Major psychiatric disorder that, in the opinion of the investigators, would impede study compliance and necessitate more intensive treatment, including major depressive disorder, bipolar disorder, posttraumatic stress disorder, panic disorder, obsessive-compulsive disorder, schizophrenia, conduct disorder, alcohol and substance abuse, and anorexia/bulimia nervosa
* Psychotherapy or structured weight loss program
* Active suicidal ideation or suicidal behavior

Ages: 12 Years to 17 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 147 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-05-26 (Actual)

PRIMARY OUTCOMES:
Depressive symptoms | 1-year
  Center for Epidemiologic Studies-Depression Scale (CES-D) total score
Insulin sensitivity | 1-year
  Whole body insulin sensitivity index estimated from 2-hour oral glucose tolerance test
Insulin secretion | 1-year
  Oral disposition index estimated from 2-hour oral glucose tolerance test

SECONDARY OUTCOMES:
Disinhibited eating | 1-year
  Emotional Eating Scale adapted for Children depression scale
Physical activity | 1-year
  Moderate-to-vigorous physical activity by accelerometer
Physical inactivity | 1-year
  Sedentary time by accelerometer
Sleep | 1-year
  Sleep duration by actigraphy
Cortisol diurnal rhythm | 1-year
  Salivary cortisol by home collection throughout the day
Daily cortisol output | 1-year
  24-hour urine cortisol

CONTACTS AND LOCATIONS:
Overall Officials: Lauren B Shomaker, PhD, Principal Investigator — Colorado State University
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shomaker LB, Gulley L, Hilkin AM, Clark E, Annameier S, Rao S, Rockette-Wagner B, Kriska A, Wright KP Jr, Stice E, Nadeau KJ, Kelsey MM. Design of a randomized controlled trial to decrease depression and improve insulin sensitivity in adolescents: Mood and INsulin sensitivity to prevent Diabetes (MIND). Contemp Clin Trials. 2018 Dec;75:19-28. doi: 10.1016/j.cct.2018.10.007. Epub 2018 Oct 17. PMID 30342256